CLINICAL TRIAL: NCT03884478
Title: PNF 2.0: A Novel, Gamified, Facebook-Integrated Personalized Normative Feedback Intervention to Reduce Alcohol Use and Negative Consequences Among Sexual Minority Women
Brief Title: A Gamified, Social Media Inspired Personalized Normative Feedback Alcohol Intervention for Sexual Minority Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R21AA025767-01A1 (NIH); 1R21AA025767-01A1 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-03-21 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Drinking; Alcohol Abuse; Alcohol; Harmful Use
Keywords: Social Norms; Personalized Normative Feedback; Sexual Minority Women
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Intervention Model Description: The web app is programmed to invite an eligible sub-sample of participants from the larger population to take part in an evaluation study during the competition's 3rd monthly round. Those who consent to participate are automatically randomized by Qualtrics Research Suite to receive 1 of 3 unique sequences of feedback (i.e., Alcohol & Stigma-Coping, Alcohol & Control, or Control topics only) during 2 intervention rounds taking place during a 6-month period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alcohol + Stigma Coping PNF (Experimental): Participants randomized to this condition will receive gamified personalized normative feedback on their alcohol use after answering questions about alcohol use and two control topics in Round 3. Then, in the very next Round of the competition (Round 4), these participants will receive gamified personalized normative feedback on their stigma coping behaviors after answering questions about their stigma coping behaviors and two control topics.
  Interventions: Behavioral: Personalized Normative Feedback
- Alcohol + Control PNF (Experimental): Participants randomized to this condition will receive gamified personalized normative feedback on their alcohol use after answering questions about alcohol use and control topics in Round 3. Then, in the very next Round of the competition (Round 4), these participants will receive gamified personalized normative feedback on one control topic (Relationships) after answering questions about their stigma coping behaviors and two control topics.
  Interventions: Behavioral: Personalized Normative Feedback
- Control PNF (Other): Participants randomized to the control arm will answer questions about the same topics as participants in the other conditions in Round 3 (Alcohol Use & Control) and Round 4 (Stigma-Coping & Control). However, in both Rounds 3 and 4 they will receive gamified PNF on control topics.
  Interventions: Behavioral: Personalized Normative Feedback

INTERVENTIONS:
Behavioral: Personalized Normative Feedback — Personalized Normative Feedback (PNF) is a popular social norms-based intervention strategy which presents individuals with a personalized, individual report designed to correct misperceived peer norms using a graphical display. Bar charts compare actual alcohol use statistics for the peer group to A) participants' estimates of peer drinking and, B) their own self-reported drinking.

SUMMARY:
Sexual minority women in the United States are more likely to drink alcohol, engage in heavy drinking, and experience alcohol-related problems than are heterosexual women. Yet, to date, no evidence-based intervention or prevention efforts have been developed to reduce alcohol consumption among female sexual minority community members. The proposed research seeks to narrow the disparity in alcohol intervention research by examining an innovative gamified personalized normative feedback (PNF) intervention to reduce drinking among sexual minority women found to frequent social media sites and overestimate norms related to peers' general alcohol use and drinking to cope with sexual minority stigma. The newly developed GANDR (Gamified Alcohol Norm Discovery and Readjustment) PNF format takes the well-established core components of a PNF alcohol intervention and delivers these components within an inviting, social media inspired, culturally-tailored online competition. This incognito intervention format is designed to be more appealing, engaging, believable, positively received, and thus effective than standard web-based PNF. The version developed for sexual minority women delivers PNF on alcohol use and stigma-coping behaviors within the context of an online game about sexual minority female stereotypes. Following two introductory rounds of play by a large cohort of sexual minority women, a sub-sample of 500 sexual minority female drinkers will be invited to participate in an evaluation study. Study participants will be randomized to receive 1 of 3 unique sequences of feedback (i.e., Alcohol & Stigma-Coping, Alcohol & Control, or Control topics only) during 2 intervention rounds taking place over a 6-month period. The randomized feedback sequences and multiple rounds of play will allow the research team to evaluate whether PNF on alcohol use reduces sexual minority women's alcohol consumption and negative consequences relative to PNF on control topics (AIM 2: H1), examine whether providing PNF on stigma-coping behaviors in addition to alcohol use further reduces alcohol use and consequences beyond alcohol PNF alone (AIM 2: H2), and identify mediators and moderators of intervention effectiveness (AIM 3).

DETAILED DESCRIPTION:
This incognito alcohol intervention is culturally tailored to appeal to heavy social media using sexual minority women residing in the US and ranging in age from 21 to 55 years. Personalized normative feedback on sexual identity and age specific descriptive drinking and stigma-coping norms are delivered to players within the context of an online competition designed to challenge sexual minority women stereotypes and increase visibility. To increase the believability of the normative statistics, players create a social media-inspired profile at registration which includes an optional photo, brief bio, links to social media accounts, and other basic information. Registered players are able to browse the profiles of others and actual norms for all topics are transparently generated by the responses of players taking part in the competition. To increase motivation and engagement, each monthly round of the competition features a point-based reward system, a leader board, and a cash prize that is awarded to the top scorer who demonstrates the greatest accuracy in perceptions of peers. To decrease defensive reactions and increase appeal, feedback topics are ostensibly selected by chance in the game with treatment PNF on alcohol use and stigma-coping behaviors delivered alongside feedback on control topics of high interest to community members (e.g., style, relationships, sex, etc.). Appeal and credibility are also gained through sponsorship and promotion of the competition by several collaborating community organizations trusted as sources for health and social information by sexual minority women.

One round of the game is played each month over a 8 month period. Players are encouraged to browse player profiles before each round and it is made clear that the goal is to grow one's score by submitting accurate guesses and strategic bets on the responses of other players in one's age and sexual identity group. Each round includes questions about 2 to 3 topics ostensibly selected by a slot machine like spinner. For each topic, players make guesses about the behaviors and experiences of other players in their age and sexual identity group, choose amounts of points to bet on these guesses being true of the group, and then contribute to actual group norms by answering parallel questions. Each round is "open" for 30 days. Once closed, players are sent a text message containing a private link at which they can see detailed results (PNF) for the round, view the leaderboard and cash prize winner, and play the next round.

Packaging this intervention as a fun, identity-relevant competition for sexual minority women rather than a transparent alcohol intervention study allows feasibility and efficacy to be evaluated simultaneously, with a high degree of ecological validity. First, 1200 sexual minority women will be recruited to take part in the online competition. No participation-based incentives will be offered to players beyond the opportunity to compete for a variable cash prize each round. Then, following two initial rounds of play, a sub-sample of 500 drinkers will be invited to take part in an incentivized evaluation study after answering alcohol use questions in Round 3. Upon consenting to participate in the evaluation study, participants will be randomized to receive 1 of 3 unique sequences of feedback (i.e., Alcohol & Stigma-Coping, Alcohol & Control, or Control only) during intervention Rounds 3 and 4. Short-term reductions in alcohol use will be assessed in Round 6 of the competition where players will be prompted to guess, bet on, and answer alcohol use and control topic questions for a second time (i.e., Replay Bonus Round; 2 month follow-up). Following all rounds of the competition, a short survey will assess the alcohol use and negative consequences of Evaluation Study participants a final time (4 month follow-up).

Feasibility analysis will examine engagement with the online competition platform and sustainability of play in the absence of traditional study participation incentives among players not involved in the Evaluation Study. Efficacy analysis will focus on study participants randomly assigned to 1 of the 3 feedback conditions in order to: 1) evaluate whether PNF on alcohol use reduces sexual minority women's alcohol consumption and negative consequences relative to PNF on control topics; 2) examine whether providing PNF on stigma-coping behaviors in addition to alcohol use further reduces alcohol use and consequences beyond alcohol PNF; and, 3) identify mediators and moderators of intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Registered for the online competition
* Accept the competition's Terms of Service & Privacy Policy
* Endorses a lesbian, bisexual, or queer female sexual identity
* Is between the ages of 21 and 55 years
* Has consumed 3 or more drinks on at least one occasion during the previous 2 months OR consumes alcohol 3 or more days per week
* Lives in North America (US or Canada)
* Does not have a partner or housemate participating
* Accepts invitation and consents to participate in the Evaluation Study

Exclusion Criteria:

* Does not register for the online competition.
* Does not accept the competition's Terms of Service & Privacy Policy
* Is younger than 21 years of age or older than 55 years of age.
* Has NOT consumed 3 or more drinks on at least one occasion during the previous 2 months AND drinks less than 3 days per week
* Lives outside of North America
* Has a partner or housemate participating
* Declines invitation
* Does not consent to participate in the Evaluation Study

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must endorse a lesbian, bisexual, or queer female sexual identity. Both the larger competition and the Evaluation Study are trans-inclusive. That is, individuals who endorse one of these sexual minority identities and presently endorse a female gender identity (regardless of whether their birth sex is female) may take part in the competition and the Evaluation Study.
Enrollment: 500 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Marymount University, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified longitudinal dataset containing data from Evaluation Study participants at will be made available to researchers 1 year after the initial publication of results. This data set will include participant demographics and outcome measures assessed at baseline (Round 3), the 2 month follow-up (Round 6), and the 4 month follow-up (a survey following the last round of the competition). A data dictionary will be provided.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year following the publication of results.
Access Criteria: The Office of Sponsored Research at Loyola Marymount University is currently working with the University's IT department to develop a data repository for the purpose of data and resource sharing. Study materials and data will be made available to the public on a secure web portal.

REFERENCES:
- [Background] Boyle SC, LaBrie JW. A Gamified, Social Media-Inspired, Web-Based Personalized Normative Feedback Alcohol Intervention for Lesbian, Bisexual, and Queer-Identified Women: Protocol for a Hybrid Trial. JMIR Res Protoc. 2021 Apr 16;10(4):e24647. doi: 10.2196/24647. PMID 33861212
- [Derived] Boyle SC, LaBrie JW, Trager BM, Costine LD. A Gamified Personalized Normative Feedback App to Reduce Drinking Among Sexual Minority Women: Randomized Controlled Trial and Feasibility Study. J Med Internet Res. 2022 May 13;24(5):e34853. doi: 10.2196/34853. PMID 35559854
- Available data/document: Study Protocol — https://www.researchprotocols.org/2021/4/e24647 — available open access at URL provided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Players learned about the broader LezParlay competition through 1 of 4 promotion strategies taking place over a 3-month period (11/15/2018 thru 2/15/2019): 1) flyers and promotional items distributed at local LBQ community events in Los Angeles; 2) targeted advertisement campaigns on HER social app, the leading LBQ dating app; 3) an advertisement in the email newsletter of Autostraddle, a popular blog for LBQ women; 4) targeted advertisement campaigns on Google, Facebook, and Instagram.
Pre-assignment Details: The 3rd round of LezParlay served as both the screening instrument and baseline assessment for the clinical trial. A total of 1337 women completed the round with the first 912 screened for clinical trial eligibility before the 500 spots in the trial were filled. One enrolled participant randomized to an arm was withdrawn prior to intervention delivery after disclosing to the research team that she had lied about her age and was actually a minor. This resulted in an N of 499.
Period: Baseline to 2 Months Post-intervention
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Started | 144 | 179 | 177
Completed | 113 | 146 | 141
Not Completed | 31 | 33 | 36
Not completed — Lost to Follow-up | 30 | 33 | 36
Not completed — Withdrawn by research team | 1 | 0 | 0
Period: Baseline to 4 Months Post-intervention
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Started | 144 | 179 | 177
Completed | 101 | 129 | 126
Not Completed | 43 | 50 | 51
Not completed — Lost to Follow-up | 42 | 50 | 51
Not completed — Withdrawn by research team | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF | Total
Number analyzed (Participants) | 143 | 179 | 177 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  years | 29.73 (7.15) | 30.37 (7.75) | 29.47 (7.03) | 29.87 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  Participants
    Female | 143 | 179 | 177 | 499
    Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  Participants
    Hispanic or Latino | 37 | 46 | 40 | 123
    Not Hispanic or Latino | 106 | 133 | 137 | 376
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant disclosed being a minor after enrollment and was withdrawn from the study
  Participants
    American Indian or Alaska Native | 4 | 5 | 4 | 13
    Asian | 6 | 16 | 17 | 39
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
    Black or African American | 19 | 25 | 26 | 70
    White | 78 | 91 | 99 | 268
    More than one race | 35 | 41 | 31 | 107
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  participants
    United States | 143 | 179 | 177 | 499
Sexual Identity [Count of Participants; unit: Participants] — Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  Participants
    Lesbian | 89 | 108 | 94 | 291
    Bisexual | 29 | 39 | 48 | 116
    Queer | 25 | 32 | 35 | 92
Interpersonal Sexual Minority Stigma Exposure [Mean (Standard Deviation); unit: units on a scale (range 0 low to 2 high)] — Two binary items assessed whether in the previous 2 months participant experienced (1) physical violence due to their sexual minority status; and, (2) verbal harassment due to their sexual minority status. Items were coded '0' No and '1' Yes and summed (scale range 0 to 2). Higher scores reflect greater recent exposure to interpersonal sexual minority stigma, which is an an outcome known to be associated with heavier drinking and alcohol-related consequences in this population. Population: 1 participant randomized to the Alcohol + Stigma Coping PNF condition disclosed being a minor after study enrollment. This participant was was withdrawn from the study and their data was excluded from analysis.
  units on a scale (range 0 low to 2 high) | .62 (.70) | .56 (.66) | .66 (.69) | .61 (.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Drinks Per Week From Baseline to the the 2 Month Follow-up
Description: At baseline and the 2 month follow-up, items assessing drinking days per week and average drinks per occasion were multiplied in order to compute number of drinks per week. These items come from the Frequency, Quantity, Max (FQM) measure. [Baer J, S. Etiology and secondary prevention of alcohol problems with young adults. Baer J S, Marlatt G A, McMahon R, J, editors. Newbury Park: Sage; 1993.] To compute the outcome, the 2 month measure of drinks per week was subtracted from the baseline measure of drinks per week such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: alcoholic drinks per week
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 113 | 146 | 141
alcoholic drinks per week | 2.75 (4.30) | 1.99 (4.57) | -.68 (5.49)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*T2 interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 2 month follow-up in the Alcohol+Coping Arm versus the Control Arm; Test type: Other; p = .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.25, Standard Error of Mean .82
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Control Arm*T2 interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 2 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p = .005, Mixed Models Analysis; Mean Difference (Final Values) = 2.31, Standard Error of Mean .77
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 2 month follow-up in the Alcohol+Coping Arm versus the Alcohol Only Arm; Test type: Other; p = .25, Mixed Models Analysis; Mean Difference (Final Values) = .94, Standard Error of Mean .82

2. Primary Outcome: Change in Number of Drinks Per Week From Baseline to the 4 Month Follow-up
Description: At baseline and the 4 month follow-up, items assessing drinking days per week and average drinks per occasion were multiplied in order to compute number of drinks per week. These items come from the Frequency, Quantity, Max (FQM) measure. [Baer J, S. Etiology and secondary prevention of alcohol problems with young adults. Baer J S, Marlatt G A, McMahon R, J, editors. Newbury Park: Sage; 1993.] To compute the outcome, the 4 month measure of drinks per week was subtracted from the baseline measure of drinks per week such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: alcoholic drinks per week
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 100 | 127 | 126
alcoholic drinks per week | 2.52 (4.68) | 1.99 (4.57) | 0.52 (5.88)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 4 month follow-up in the Alcohol+Coping Arm versus the Control Arm; Test type: Other; p = .025, Mixed Models Analysis; Mean Difference (Final Values) = 1.90, Standard Error of Mean .84
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*T2 interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 4 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p = .11, Mixed Models Analysis; Mean Difference (Final Values) = 1.24, Standard Error of Mean .79
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 4 month follow-up in the Alcohol+Coping Arm versus the Alcohol+Control Arm; Test type: Other; p = .66, Mixed Models Analysis; Mean Difference (Final Values) = 0.66, Standard Error of Mean .84

3. Primary Outcome: Change in Peak Drinks on One Occasion From Baseline to the 2 Months Follow-up
Description: At baseline and the 2 month follow-up, an item assessing the number of maximum drinks on one occasion from the Frequency, Quantity, Max (FQM) measure was used to assess peak drinks on one occasion over the past 30 days. [Baer J, S. Etiology and secondary prevention of alcohol problems with young adults. Baer J S, Marlatt G A, McMahon R, J, editors. Newbury Park: Sage; 1993.] To compute the outcome, the 2 month measure of peak drinks was subtracted from the baseline measure of peak drinks such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: alcoholic drinks
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 143 | 179 | 177
alcoholic drinks | 1.49 (1.78) | 1.42 (1.86) | -.18 (1.92)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in peak drinks from baseline to the 2 month follow-up in the Alcohol+Coping Arm versus the Control Arm; Test type: Other; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 1.51, Standard Error of Mean .25
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on peak drinks. To probe the significant Alcohol+Control Arm*Time interaction, a Tukey post-hoc test examined the change in peak drinks at the 2 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 1.48, Standard Error of Mean .23
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on peak drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in peak drinks at the 2 month follow-up in the Alcohol+Coping Arm versus the Alcohol+Control Arm; Test type: Other; p = .88, Mixed Models Analysis; Mean Difference (Final Values) = .04, Standard Error of Mean .25

4. Primary Outcome: Change in Peak Drinks on One Occasion From Baseline to the 4 Month Follow-up
Description: At baseline and the 4 month follow-up, an item assessing the number of maximum drinks on one occasion from the Frequency, Quantity, Max (FQM) measure was used to assess peak drinks on one occasion over the past 30 days. [Baer J, S. Etiology and secondary prevention of alcohol problems with young adults. Baer J S, Marlatt G A, McMahon R, J, editors. Newbury Park: Sage; 1993.] To compute the outcome, the 4 month measure of peak drinks was subtracted from the baseline measure of peak drinks such that a positive value indicates a decrease in consumption during this period and a negative value indicates an increase in consumption during this period.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: alcoholic drinks
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 113 | 146 | 126
alcoholic drinks | .82 (1.71) | .61 (1.46) | .08 (2.06)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .03, Mixed Models Analysis; Mean Difference (Final Values) = .55, Standard Error of Mean .26
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on peak drinks. To probe the significant Alcohol+Control Arm*Time interaction, a Tukey post-hoc test examined the change in weekly drinks from baseline to the 4 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p = .059, Mixed Models Analysis; Mean Difference (Final Values) = .46, Standard Error of Mean .24
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on weekly drinks. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in peak drinks from baseline to the 4 month follow-up in the Alcohol+Coping Arm versus the Alcohol+Control Arm; Test type: Other; p = .71, Mixed Models Analysis; Mean Difference (Final Values) = .10, Standard Error of Mean .26

5. Primary Outcome: Change in Number of Negative Alcohol-related Consequences From Baseline to the 2 Month Follow-up
Description: At baseline and the 2 month follow-up, a single item assessed the number of negative alcohol-related consequences experienced out of a list of 8 common negative alcohol-related consequences. This item is adapted from Riley BB, Hughes TL, Wilsnack SC. Validating a hazardous drinking index in a sample of sexual minority women: Reliability, validity, and predictive accuracy. Substance Use and Misuse. 2017;52(1):43-51. doi: 10.1080/10826084.2016.1214150.] To compute the outcome, the 2 month measure of negative consequences was subtracted from the baseline measure of negative consequences such that a positive value indicates a decrease in consequences during this period and a negative value indicates an increase in consequences during this period.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: negative consequences
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 113 | 146 | 141
negative consequences | .23 (1.82) | .25 (1.56) | -.76 (1.68)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 2 month follow-up in the Alcohol+Coping Arm versus the Control Arm; Test type: Other; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = .86, Standard Error of Mean .20
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Control Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 2 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = .83, Standard Error of Mean .18
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 2 month follow-up in the Alcohol+Coping Arm versus the Alcohol+Control Arm; Test type: Other; p = .87, Mixed Models Analysis; Mean Difference (Final Values) = .03, Standard Error of Mean .19

6. Primary Outcome: Change in Number of Negative Alcohol-related Consequences From Baseline to the 4 Month Follow-up
Description: At baseline and the 4 month follow-up, a single item assessed the number of negative alcohol-related consequences experienced out of a list of 8 common negative alcohol-related consequences. This item is adapted from Riley BB, Hughes TL, Wilsnack SC. Validating a hazardous drinking index in a sample of sexual minority women: Reliability, validity, and predictive accuracy. Substance Use and Misuse. 2017;52(1):43-51. doi: 10.1080/10826084.2016.1214150.] To compute the outcome, the 4 month measure of negative consequences was subtracted from the baseline measure of negative consequences such that a positive value indicates a decrease in consequences during this period and a negative value indicates an increase in consequences during this period.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: negative consequences
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
Number analyzed (Participants) | 100 | 127 | 126
negative consequences | .34 (1.55) | .21 (1.56) | -.67 (1.59)
Statistical Analysis 1: Comparison: Alcohol + Stigma Coping PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 4 month follow-up in the Alcohol+Coping Arm versus the Control Arm; Test type: Other; p < .001, Mixed Models Analysis; Median Difference (Final Values) = .86, Standard Error of Mean .20
Statistical Analysis 2: Comparison: Alcohol + Control PNF vs Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Control Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 4 month follow-up in the Alcohol+Control Arm versus the Control Arm; Test type: Other; p = .002, Mixed Models Analysis; Mean Difference (Final Values) = .70, Standard Error of Mean .19
Statistical Analysis 3: Comparison: Alcohol + Stigma Coping PNF vs Alcohol + Control PNF; As detailed in the statistical analysis plan, a multi-level model which held constant participant age, race, ethnicity, relationship status, sexual identity, and sexual minority interpersonal stigma exposure in examining Time*Arm interactions on negative consequences. To probe the significant Alcohol+Coping Arm*Time interaction, a Tukey post-hoc test examined the change in negative consequences from baseline to the 4 month follow-up in the Alcohol+Coping Arm versus the Alcohol+Control Arm; Test type: Other; p = .43, Mixed Models Analysis; Mean Difference (Final Values) = .15, Standard Error of Mean .20

ADVERSE EVENTS:
Time Frame: 8 months
Description: Participants were provided contact information (phone, email, and in-app direct message address) at which they were asked to report any negative outcomes they experienced over the competition and study period.
Arm/Group | Alcohol + Stigma Coping PNF | Alcohol + Control PNF | Control PNF
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/179 | 0/177
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/179 | 0/177
Other Adverse Events (participants affected / at risk) | 0/143 | 0/179 | 0/177

LIMITATIONS AND CAVEATS:
No limitations. However, in hindsight it would have been ideal to have included an assessment only control arm, which would have allowed us to evaluate app use effects beyond the PNF received.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03884478/Prot_003.pdf
  • Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03884478/SAP_004.pdf
  • Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03884478/ICF_002.pdf